CLINICAL TRIAL: NCT04683159
Title: The Effect of Brimonidine Tartrate on Subconjunctival Hemorrhage During Pterygium Surgery
Brief Title: Brimonidine Tartrate for Pterygium Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uptown Eye Specialists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Red Eye 2.0
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Pterygium; Subconjunctival Hemorrhage
Keywords: Brimonidine tartrate; Pterygium surgery; Subconjunctival hemorrhage
MeSH Terms: conditions — Pterygium | interventions — Brimonidine Tartrate

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups (control, brimonidine 0.15%, or brimonindine 0.025%), running in parallel.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeon (care provider/investigator) will be masked to the intervention at the time of operation and during follow-ups (day 0, week 1, month 1). Outcomes assessor will be blinded to the investigation when quantifying degree of hemorrhage
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): No intervention, only routine pre-operative drops
- Brimonidine 0.15% (Experimental): Routine pre-operative drops + 1 drop of brimonidine tartrate 0.15% in the operating eye
  Interventions: Drug: Brimonidine Tartrate 0.15% Oph Soln
- Brimonidine 0.025% (Experimental): Routine pre-operative drops + 1 drop of brimonidine tartrate 0.025% in the operating eye
  Interventions: Drug: Brimonidine Tartrate 0.025% Oph Soln

INTERVENTIONS:
Drug: Brimonidine Tartrate 0.15% Oph Soln — 1 drop of brimonidine 0.15% (~0.05mL) 15 minutes prior to surgery
  Other Names: Alphagan-P
  Arms: Brimonidine 0.15%
Drug: Brimonidine Tartrate 0.025% Oph Soln — 1 drop of brimonidine 0.025% (~0.05mL) 15 minutes prior to surgery
  Other Names: Lumify
  Arms: Brimonidine 0.025%

SUMMARY:
Pterygium excision and conjunctival autograft surgery is commonly done to treat pterygiums. Excessive bleeding during the procedure creates a challenging operating field, prolongs surgery time, and prolongs healing.

Brimonidine tartrate has a vasoconstrictive effect, which helps to reduce the amount of blood flow and hyperemia to the eye. Preoperative use of brimonidine has been shown to decrease subconjunctival hemorrhage during procedures such as cataract surgery, laser assisted in situ keratomileusis, strabismus surgery, and intravitreal injections. The focus of this study is to assess the effect of preoperative application of brimonidine tartrate 0.15% (Alphagan) and 0.025% (Lumify) on reducing hemorrhage during pterygium excision and conjunctival autograft surgery.

DETAILED DESCRIPTION:
During pterygium excision and conjunctival autograft surgery, incision into the conjunctiva of the operated eye causes a significant amount of subconjunctival hemorrhage. Brimonidine-tartrate is a selective alpha-2-adrenergic agonist. The 0.15% concentration (Alphagan) is commonly used to treat glaucoma, while the 0.025% (Lumify) is an over-the-counter drop used for its vasoconstrictive anti-hyperemia effect. Brimonidine 0.15% has been evaluated in other studies to reduce bleeding in LASIK, cataract surgery, strabismus surgery, as well as intravitreal injections. In these mentioned clinical trials, brimonidine was found to safely reduce subconjunctival hemorrhage intraoperatively and hyperemia postoperatively. Interestingly, prophylactic topical brimonidine was found to increase risk of early flap slippage in LASIK due to molecular interference with flap stabilization. Because creation of a flap is not a component of pterygium surgery, preoperative brimonidine does not interfere with healing.

A recent study by Ucar et al. has validated the use of preoperative brimonidine 0.15% for conjunctival whitening prior to pterygium surgery, allowing for minimized hyperemia and reduced surgical duration (Ucar, 2020). However, the long-term clinical outcomes, and efficacy of brimonidine 0.025% has yet to be examined. This study aims to further examine the comparative efficacy of preoperative brimonidine at different concentrations to reduce subconjunctival hemorrhage during pterygium surgery.

Potential side effects of topical application of brimonidine eye drop may include blurred or loss of vision, burning, dry, or itching eyes, discharge or excessive tearing, disturbed color perception, double vision, halos around lights, headache, itching of the eye, night blindness, photophobia, redness of the eye or inner lining of the eyelid, swelling of the eyelid, tearing of the eye, tunnel vision. Side effects of this medication are self-limited, and reversible after the medication is stopped.

The risk of this study to the subject is negligible as the standard surgical procedure will be followed. This trial will be conducted in compliance with the protocol, GCP, and the applicable regulatory requirement as set by William Osler Health System Ethics Review Board.

ELIGIBILITY:
Inclusion Criteria:

* All patients over age 18 who are scheduled for pterygium surgery who have provided informed consent, in accordance with application regulations and guidelines

Exclusion Criteria:

* Patients who are on anticoagulation or antiplatelet therapy
* Patients on monoamine oxidase (MOA) inhibitor therapy
* Patients who have undergone any conjunctival surgery in the past
* Any complication during pterygium excision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Subconjunctival hemorrhage grading | Post-operative Day 0 (30 minutes following operation)
  Subconjunctival hemorrhage grading of images at POD0, POW1, and POM1 will be done as follows: a score of 1-4 for the number of quadrants involved, and a score of 1-4 for the amount of involvement in the quadrant (1 = 0-25% coverage, 2 = 26-50% coverage, 3 = 51-75% coverage, 4 = 76-100% coverage). A total maximum score of 16 may be given, with 0 indicating no subconjunctival hemorrhage present. This grading algorithm is adapted from previously published methods (Munoz 2009, Hong 2007, Norden 2002). Grading will be done by an independent reviewer blinded to the randomization of participants.
Subconjunctival hemorrhage grading | Post-operative Week 1
  Subconjunctival hemorrhage grading of images will be done as follows: a score of 1-4 for the number of quadrants involved, and a score of 1-4 for the amount of involvement in the quadrant (1 = 0-25% coverage, 2 = 26-50% coverage, 3 = 51-75% coverage, 4 = 76-100% coverage). A total maximum score of 16 may be given, with 0 indicating no subconjunctival hemorrhage present. This grading algorithm is adapted from previously published methods (Munoz 2009, Hong 2007, Norden 2002). Grading will be done by an independent reviewer blinded to the randomization of participants.
Subconjunctival hemorrhage grading | Post-operative Month 1 (4 weeks)
  Subconjunctival hemorrhage grading of images will be done as follows: a score of 1-4 for the number of quadrants involved, and a score of 1-4 for the amount of involvement in the quadrant (1 = 0-25% coverage, 2 = 26-50% coverage, 3 = 51-75% coverage, 4 = 76-100% coverage). A total maximum score of 16 may be given, with 0 indicating no subconjunctival hemorrhage present. This grading algorithm is adapted from previously published methods (Munoz 2009, Hong 2007, Norden 2002). Grading will be done by an independent reviewer blinded to the randomization of participants.

SECONDARY OUTCOMES:
Hyperemia | Baseline
  Hyperemia will be quantified in the same manner as Ucar et al. (Ucar, 2020). Vessels on the images converted to black and white with Adobe Photoshop - vessels will be converted to black, while the rest of the sclera will be white. ImageJ (public domain software) will then be used to quantify the number of black pixels (vessels). Hyperemia will be reported as the number of black pixels per image.
Hyperemia | Post-drop (5 minutes after administration)
  Hyperemia will be quantified in the same manner as Ucar et al. (Ucar, 2020). Vessels on the images converted to black and white with Adobe Photoshop - vessels will be converted to black, while the rest of the sclera will be white. ImageJ (public domain software) will then be used to quantify the number of black pixels (vessels). Hyperemia will be reported as the number of black pixels per image.
Hyperemia | Post-operative day 0 (30 minutes after surgery)
  Hyperemia will be quantified in the same manner as Ucar et al. (Ucar, 2020). Vessels on the images converted to black and white with Adobe Photoshop - vessels will be converted to black, while the rest of the sclera will be white. ImageJ (public domain software) will then be used to quantify the number of black pixels (vessels). Hyperemia will be reported as the number of black pixels per image.
Hyperemia | Post-operative week 1
  Hyperemia will be quantified in the same manner as Ucar et al. (Ucar, 2020). Vessels on the images converted to black and white with Adobe Photoshop - vessels will be converted to black, while the rest of the sclera will be white. ImageJ (public domain software) will then be used to quantify the number of black pixels (vessels). Hyperemia will be reported as the number of black pixels per image.
Hyperemia | Post-operative month 1
  Hyperemia will be quantified in the same manner as Ucar et al. (Ucar, 2020). Vessels on the images converted to black and white with Adobe Photoshop - vessels will be converted to black, while the rest of the sclera will be white. ImageJ (public domain software) will then be used to quantify the number of black pixels (vessels). Hyperemia will be reported as the number of black pixels per image.
Duration of operation | During surgery
  The length of time it takes the pterygium operation
Visual Acuity | Baseline
  logMAR visual acuity
Visual Acuity | Post-operative week 1
  logMAR visual acuity
Visual Acuity | Post-operative month 1
  logMAR visual acuity
Steroid usage | Post-operative week 1
  Duration & frequency of steroid usage
Steroid usage | Post-operative month 1
  Duration & frequency of steroid usage

CONTACTS AND LOCATIONS:
Overall Officials: Eric Tam, MD, Principal Investigator — Uptown Eye Specialists

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desco MC, Navea A, Ferrer E, Menezo JL. Effect of prophylactic brimonidine on bleeding complications after cataract surgery. Eur J Ophthalmol. 2005 Mar-Apr;15(2):228-32. doi: 10.1177/112067210501500209. PMID 15812765
- [Background] Hong S, Kim CY, Seong GJ, Han SH. Effect of prophylactic brimonidine instillation on bleeding during strabismus surgery in adults. Am J Ophthalmol. 2007 Sep;144(3):469-70. doi: 10.1016/j.ajo.2007.04.038. PMID 17765438
- [Background] Kim CS, Nam KY, Kim JY. Effect of prophylactic topical brimonidine (0.15%) administration on the development of subconjunctival hemorrhage after intravitreal injection. Retina. 2011 Feb;31(2):389-92. doi: 10.1097/IAE.0b013e3181eef28e. PMID 20890238
- [Background] Munoz G, Albarran-Diego C, Sakla HF, Javaloy J. Increased risk for flap dislocation with perioperative brimonidine use in femtosecond laser in situ keratomileusis. J Cataract Refract Surg. 2009 Aug;35(8):1338-42. doi: 10.1016/j.jcrs.2009.03.029. PMID 19631117
- [Background] Norden RA. Effect of prophylactic brimonidine on bleeding complications and flap adherence after laser in situ keratomileusis. J Refract Surg. 2002 Jul-Aug;18(4):468-71. doi: 10.3928/1081-597X-20020701-10. PMID 12160159
- [Background] Ucar F, Cetinkaya S. The Results of Preoperative Topical Brimonidine Usage in Pterygium Surgery. J Ocul Pharmacol Ther. 2020 May;36(4):234-237. doi: 10.1089/jop.2019.0085. Epub 2020 Feb 27. PMID 32105500